CLINICAL TRIAL: NCT05962034
Title: The Role of Thomboxane A2 and it's Receptor in Vascular Regulation in Women With Endometriosis
Brief Title: Thromboxane Function in Women With Endometriosis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Lacy Alexander, Professor of Kinesiology, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 21851
Record Dates: First submitted 2023-06-30; First posted 2023-07-27 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Endometriosis
Keywords: Endometriosis; Aspirin
MeSH Terms: conditions — Endometriosis | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin (Experimental): one dose of aspirin
  Interventions: Drug: Aspirin
- Placebo (Placebo Comparator): Placebo pill
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Aspirin — 650 mg aspirin (Acetylsalicylic acid)
  Arms: Aspirin
Other: Placebo — placebo capsule
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to compare neurovascular regulation in women with endometriosis and healthy women. The main questions it aims to answer are:

* Do women with endometriosis have greater blood pressure and pain responses to a stimulus than healthy women?
* Do women with endometriosis have greater platelet activity than healthy women?

Participants will take aspirin and/or placebo and will:

* perform hand grip exercise and cold pressor tests
* undergo iontophoresis and blood draw

Researchers will compare women with and without endometriosis to see if there is a difference in neurovascular regulation.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of death worldwide. Endometriosis is an independent risk factor for CVD that affects an estimated one in ten women in the world. Endometriosis is a gynecologic condition characterized by invasive extrauterine endometriotic lesions, chronic pain, and systemic inflammation. The expression of thromboxane A2 (TxA2), a product of the inflammatory cyclooxygenase pathway, is upregulated in endometriotic lesions. In the vasculature, TxA2 blocks vasodilation, and induces vasoconstriction. TxA2 diffuses across the innermost layer of cells in the blood vessels, the endothelium, to act directly on its receptors in the vascular smooth muscle. It also inhibits endothelial nitric oxide synthase, thereby decreasing nitric oxide (NO)-mediated vasodilation --endothelial dysfunction which is regarded as a critical early event in the development of atherosclerosis and overt cardiovascular disease. Women with endometriosis demonstrate marked endothelial dysfunction compared with healthy controls, but the potential role of TxA2 and its receptors (TP) in this dysfunction have not been investigated. Furthermore, TP play a key role in sensitizing the sensory afferent nerve fibers in pre-clinical models of cardiovascular disease, leading to an exaggerated blood pressure responses to sympathoexcitatory maneuvers including the exercise pressor reflex. The exercise pressor reflex is the reflex increase in blood pressure in response to the mechanical and metabolic stimuli of exercise. The exaggeration of this reflex response is a strong predictor of major adverse cardiovascular events in cardiovascular disease patients. However, the reflex response to sympathoexcitatory maneuvers has not been characterized in women with endometriosis. Furthermore, TxA2 is a key component in the clotting cascade. An increased production of TxA2 in the platelet cells of women with endometriosis indicates altered platelet function. However, platelet activity in women with endometriosis has not been characterized.

ELIGIBILITY:
Inclusion Criteria:

* Born with a uterus
* 18-45 years old
* With and without endometriosis

Exclusion Criteria:

* Currently pregnant or breastfeeding
* Diagnosed cardiovascular disease
* BMI over 35
* Nicotine use (e.g., smoking, chewing tobacco, vaping, etc.)
* Currently using hormone replacement therapy (or have used within previous 6 months)
* Known skin allergies or current rash, skin disease, disorders of pigmentation
* Diabetes
* Renal disease, renal artery stenosis, renal impairment
* Liver disease
* Stage II Hypertension (blood pressure >140/>90 mmHg)
* Hypotension (blood pressure < 90/60 mmHg)
* Raynaud's syndrome
* Any current medications which could conceivably alter cardiovascular responses (e.g. antihypertension medication, diuretic, digoxin)
* Allergy or hypersensitivity to investigational agents
* Immunosuppressed/immunocompromised

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
blood pressure | 1 day
  change in blood pressure from baseline to maximum
heart rate | 1 day
  change in heart rate from baseline to maximum
pain scale | 1 day
  pain scale rating in response to testing
skin blood flow | 1 day
  change in skin blood flow from baseline to maximum

CONTACTS AND LOCATIONS:
Locations (1):
- Noll Laboratory, University Park, Pennsylvania, United States